CLINICAL TRIAL: NCT00426816
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Effects of SB-649868 (10, 30 mg and 60 mg) on Sleep Continuity, PSG Sleep Recordings, Subjective Sleep Assessment, and Daytime Cognitive Function in Subjects With Primary Insomnia
Brief Title: To Evaluate The Effects Of SB-649868 (10, 30 Mg And 60 Mg) On Subjects With Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OXS107714
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: primary insomnia; PSG sleep recordings; daytime cognitive function; Insomnia; SB-649868
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Crossover population (Experimental): All study population receive placebo and doses of SB-649868 at 10mg, 30mg and 60mg in a crossover desing
  Interventions: Drug: SB-649868; Drug: Placebo

INTERVENTIONS:
Drug: SB-649868 — Active compound at doses of 10mg, 30mg and 60mg
Drug: Placebo — Placebo to match SB-649868

SUMMARY:
This study to evaluate the effects of SB-649868 (10, 30 mg and 60 mg) on sleep continuity, PSG sleep recordings, subjective sleep assessment, and daytime cognitive function in subjects with primary insomnia

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-64 years of age (inclusive),
* Diagnosis of primary insomnia who have had symptoms for at least three months.

Exclusion Criteria:

* Any clinically significant unstable medical or surgical condition (treated or untreated).
* Any history of a clinically significant abnormality of the neurological system (including cognitive disorders or significant head injury) or any history of seizure (including febrile seizure).

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time (TST), Latency to Persistent Sleep (LPS) and Wake time after sleep onset (WASO) derived from polysomongraphic (PSG) recording. | 9 weeks
  Statistical paramaters of sleep measured by analysis of Polysomnography during night section of subject visit. Measured for one night during each 4 study visits and twice at screening. All visits will take in total approximately 9 weeks from screening to follow-up.

SECONDARY OUTCOMES:
Objective PSG measures of sleep continuity including: wake during sleep (WDS), wake after sleep (WAS), and number of awakenings during sleep. Objective PSG measures of sleep structure | 9 weeks
  Real time Polysomnography technique using combination of EEG, ECG, EOG and EMG to collect data on physiological cleep activity. Data/graphs are collected and analysed post sleep. Measured for one night during each 4 study visits and twice at screening. All visits will take in total approximately 9 weeks from screening to follow-up.
Objective PSG measures of sleep structure: Non-REM sleep time, Slow-Wave Sleep (SWS) time (stage 3 and 4), Stage 2 non-REM sleep time; REM sleep time, REM activity, REM density. | 9 weeks
  Real time Polysomnography technique using combination of EEG, ECG, EOG and EMG to collect data on physiological cleep activity. Data/graphs are collected and analysed post sleep. Measured for one night during each 4 study visits and twice at screening. All visits will take in total approximately 9 weeks from screening to follow-up.
Spectral analysis of EEG | 9 weeks
  Collected as part of PSG. Graph spectra can be quantitatively analysed to assess electrical activity in the brain. Measured for one night during each 4 study visits and twice at screening. All visits will take in total approximately 9 weeks from screening to follow-up.
Subjective Post-Sleep Questionnaire: TST, WASO, SOL, number of awakenings, and sleep quality (SQ) to be applied on each morning following PSG recording. | 9 weeks
  Subject answers sleep quality questionnaires after night of sleep during the visit. Measured for each morning after each 4 study night visits and twice at screening. All visits will take in total approximately 9 weeks from screening to follow-up.
Daytime cognitive function data on the morning following dosing, including tests of alertness, memory, attention and fine motor control (i.e. Romberg, VAS for sleepiness/alertness, DSST, and immediate and delayed word recall). | 9 weeks
  Measurements of insomnia effects on daytime regular functions
HVLT-R (verbal memory tests), TST, SOL, SQ, WAS and number of awakenings measured with the Post-Sleep Questionnaire score collected on specified mornings at home during the 3-day period following each 2-night PSG sessions. | 9 weeks
  Further questionnaires answered after each visit regarding sleep quality. Measured during night and day sections at each visit depending on the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Germany (8):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin, State of Berlin